CLINICAL TRIAL: NCT01129869
Title: Research Participant Perception of Care Project: Part II: Fielding and Validation of the Research Participant Perception Survey Derived From Focus Group-Identified Key Dimensions of the Research Participant Experience
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999910127; 10-CC-N127
Record Dates: First submitted 2010-05-22; First posted 2010-05-25 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-02-01

CONDITIONS: Participation Satisfaction
Keywords: Survey; Perception; Perception of Clinical Research Participation; Research Participant Perception

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Understanding participants experiences as research volunteers is critical to improving the effectiveness of human participant protection programs and strengthening public trust in clinical research. Historically, studies that evaluate participants comprehension of the informed consent document or evaluate the informed consent process have only indirectly measured the quality of a participant s experience.
* Few studies have assessed the nature, quality and efficiency of the entire clinical research process from the participant s perspective. To address this need, researchers have developed a Clinical Research Participant Perception Survey to evaluate participants overall perceptions of clinical research.

Objectives:

- To validate the Research Participant Perception Survey questionnaire and revise it accordingly to produce a questionnaire that other researchers can use.

Eligibility:

- Individuals at least 18 years of age who have participated in at least one research protocol within the past 2 years. Participation may be completed or ongoing.

Design:

* Eligible participants will receive a survey by mail and will be asked to complete it and return it in the stamped envelope provided.
* The survey will ask questions about the research protocol process, including participants positive and negative experiences of participating in the research protocol....

DETAILED DESCRIPTION:
Understanding participants experiences as research volunteers is critical to improving the effectiveness of human participant protection programs, and strengthening the public trust in the clinical research enterprise. Institutional Review Boards, investigators and regulators have few tools, little direct information, and no validated outcome measures in this regard. Yet, to operate rationally, IRBs and investigations need not only data on local performance, but also the critical ability to benchmark among peers and identify best practices. Historically, studies evaluating participant s comprehension of the informed consent document or evaluating the informed consent process have served, at best, as indirect measures of the quality of the participant s experience, focusing primarily on the readability of text and institutional process. Few if any studies have assessed the nature, quality and efficiency of the entire clinical research process from the participant s perspective, nor produced results that are actionable and relevant to the research participant experience.

This study is the second phase of a two-part study designed to directly measure research participants perceptions of the clinical research process as defined by what research participants themselves have articulated in focus groups as the relevant aspects of their clinical research experience. In the first phase of the project, from May 2008- November 2008, 89 research volunteers and 29 research professionals from eight academic research institutions were enrolled into 18 focus groups to assess the key dimensions of the research experience. Using qualitative research methods, the main themes of the research participant experience were extracted from the analysis of the transcripts of those focus groups and a draft survey was constructed. The current protocol describes the fielding and validation of the Research Participant Perception Survey instrument in 15 academic research institutions across the Clinical and Translational Science Awards (CTSA) consortium. The scope of the fielding and validation study is enhanced by the support of a CTSA Administrative Supplement which facilitated the increase of the number of participating centers from 9 to 15 institutions, and enlarges the sample size of completed surveys from 3600 to 5400 completed participant surveys (based on 340 completed surveys/institution for 95% confidence intervals.) Based on prior experience of 45% return rates, it is estimated that 10,000 surveys will be deployed across the 15 institutions in order to obtain the targeted 5400 completed surveys.

Leveraging the hospital survey expertise of our colleagues at NRC Picker, the fielding of the draft survey instrument is designed to validate the instrument and to attain highly relevant, actionable process and outcome measures. Survey data may be used for benchmarking and to assist centers in identifying best practices to offer the consortium. Center-specific survey data may be used to improve the clinical research participant experience, enhance public trust, and to strengthen the clinical research enterprise. Information regarding the processes of study design and implementation during this intra-consortium collaboration will also be derived to streamline and improve such collaborations in the future.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 years or older.

Subject has been a participant in at least one research protocol within the past two years, as recorded by the participating center (participation may be over, or ongoing).

Ability to give consent/permission; this requirement may waived if pror permission for future contact is in place, or IRB waiver of written consent has been granted.

EXCLUSION CRITERIA:

Individuals whose research participation contact is limited to being the parent of a pediatric research participant.

Individuals who are legally authorized representatives for participants.

Individuals who were eligible for but did not enroll in a research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2010-05-13; Study Completion 2018-02-01

PRIMARY OUTCOMES:
To validate the Research Participant Perception Survey instrument and revise accordingly to produce and instrument for broader application.

SECONDARY OUTCOMES:
To collect and disseminate data from the results of the multi-center fielding of the survey, for the purposes of benchmarking and performance improvement in the conduct of clinical translational research/

CONTACTS AND LOCATIONS:
Overall Officials: David K Henderson, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States